CLINICAL TRIAL: NCT01149486
Title: A Relative Bioavailability Study of 100/25 mg Losartan Potassium/Hydrochlorothiazide Tablets Under Fasting Conditions
Brief Title: Losartan Potassium/Hydrochlorothiazide 100/25 mg Tablets in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R04-080
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — hydrochlorothiazide, losartan drug combination; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic Test Product (Experimental): Losartan potassium/Hydrochlorothiazide 100/25 mg Tablets
  Interventions: Drug: Losartan potassium/Hydrochlorothiazide
- Reference Listed Drug (Active Comparator): Hyzaar® 100/25 mg Tablets
  Interventions: Drug: Hyzaar®

INTERVENTIONS:
Drug: Losartan potassium/Hydrochlorothiazide — 100/25 mg Tablets
  Arms: Generic Test Product
Drug: Hyzaar® — 100/25 mg Tablets
  Other Names: Losartan potassium/Hydrochlorothiazide (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The object of this study was to compare the relative bioavailability (rate and extent of absorption) of 100/25 mg Losartan potassium/Hydrochlorothiazide Tablets manufactured by Teva Pharmaceutical Industries Ltd. and distributed by Teva Pharmaceuticals USA with that of Hyzaar® 100/25 mg Tablets distributed by Merck & Co., Inc. following a single oral dose (1 x 100/25 mg tablet) in healthy adult subjects administered under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, 18-45 years of age (inclusive).
* Body mass index should be less than or equal to 30
* Screening procedures completed within 28 days prior to dosing.
* If female and:

  * of child bearing potential, is practicing an acceptable barrier method of birth control for the duration of the study
  * is postmenopausal for at least 1 year
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* Subjects with a recent history of drug or alcohol abuse or addiction.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a positive hepatitis B surface antigen screen, a positive hepatitis C antibody screen, or a reactive HIV antibody screen.
* Subjects demonstrating a positive drug abuse screen when screened for the study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breastfeeding.
* Subjects who have used implanted or injected hormonal contraceptives anytime during the 180 days prior to study dosing or hormonal contraceptives within 14 days of dosing will not be allowed to participate.
* Subjects with a history of allergic response(s) to losartan, hydrochlorothiazide or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to dosing (as determined by the clinical investigators).
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to dosing.
* Subjects who have used tobacco products within 90 days of Period 1 dose administration.
* Subjects who report donating greater than 150 mL of blood within 14 days prior to dosing.
* Subjects who report receiving any investigational drug within 28 days prior to dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet within the 28 days prior to dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan/HCTZ (Test) First: 100/25 mg Losartan potassium/Hydrochlorothiazide Tablets test product dosed in first period followed by 100/25 mg Hyzaar® Tablets reference product dosed in the second period.
- Hyzaar® (Reference) First: 100/25 mg Hyzaar® Tablets reference product dosed in first period followed by 100/25 mg Losartan potassium/Hydrochlorothiazide Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout of 7 Days
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 1 | 1 | 2
  Black | 0 | 1 | 1
  Caucasian | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Losartan(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Losartan Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Losartan/HCTZ (Test): 100/25 mg Losartan potassium/Hydrochlorothiazide Tablets test product dosed in either period.
- Hyzaar® (Reference): 100/25 mg Hyzaar® Tablets reference product dosed in either period.
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng/mL | 509.63 (314.75) | 538.11 (298.89)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 93.45, 90% CI 2-sided [80.20 to 108.88] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Losartan(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Losartan AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 866.88 (366.15) | 865.00 (362.86)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.45, 90% CI 2-sided [93.15 to 106.18] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Losartan(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Losartan AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 880.15 (368.58) | 877.99 (362.75)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.4, 90% CI 2-sided [93.10 to 106.12] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Hydroclorothiazide(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Hydrochlorothiazide Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng/mL | 177.63 (48.09) | 161.56 (53.75)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 111.62, 90% CI 2-sided [101.47 to 122.79] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Hydrochlorothiazide(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Hydrochlorothiazide AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 1057.58 (231.26) | 1001.54 (236.00)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 105.8, 90% CI 2-sided [99.58 to 112.41] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Hydrochlorothiazide(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Hydrochlorothiazide AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 1087.64 (240.82) | 1030.73 (238.96)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 105.55, 90% CI 2-sided [99.64 to 111.82] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Cmax of Losartan Carboxy Acid(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for the metabolite Losartan Carboxy Acid.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng/mL | 726.85 (210.78) | 675.54 (197.25)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 106.78, 90% CI 2-sided [98.96 to 115.23] — This analysis was for informational purposes only and was not used to establish bioequivalence

8. Secondary Outcome: AUC0-t of Losartan Carboxy Acid(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for the metabolite Losartan Carboxy Acid.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 4236.78 (1176.34) | 4117.07 (1087.67)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.37, 90% CI 2-sided [98.75 to 106.14] — This analysis was for informational purposes only and was not used to establish bioequivalence

9. Secondary Outcome: AUC0-inf of Losartan Carboxy Acid(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for the metabolite Losartan Carboxy Acid.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 19 | 19
ng*h/mL | 4281.32 (1182.77) | 4164.62 (1096.64)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.3, 90% CI 2-sided [98.72 to 106.01] — This analysis was for informational purposes only and was not used to establish bioequivalence

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan/HCTZ (Test) (N=20) | Hyzaar® (Reference) (N=20)
Headache (General disorders) | 3 (3) | 3 (3)
Pharyngitis (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (2)
Sweaty (General disorders) | 1 (1) | 0 (0)
Purpura (General disorders) | 1 (1) | 0 (0)
Leg Muscles Tight (General disorders) | 0 (0) | 1 (1)
Cut Forearm (General disorders) | 0 (0) | 1 (1)
Fell (General disorders) | 0 (0) | 1 (1)
Confussion (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.